CLINICAL TRIAL: NCT05825729
Title: Diagnostic Efficacy Of 3 Endoscopic Ultrasound-Guided Fine Needle Biopsy Techniques In Solid Masses: A Randomized Clinical Trial
Brief Title: Diagnostic Efficacy Of 3 EUS-FNB Techniques
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Insular Gran Canaria (Other)
Responsible Party: Principal Investigator, Guillermo Pérez Aguado, Principal Investigator, Hospital Universitario Insular Gran Canaria
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: TEC-EUS
Record Dates: First submitted 2023-03-22; First posted 2023-04-24 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Efficacy, Self
Keywords: endoscopic ultrasound; solid masses; fine needle biopsy

STUDY DESIGN:
Intervention Model Description: Multicentric, randomized comparative clinical trial, single-blind and crossover.
Who Masked: Participant, Outcomes Assessor
Masking Description: The anatomo-pathologist who will analyze the samples obtained in each of the techniques will not know their order or which one he/she will be analyzing. The participants will also be blind to the same.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- ABC (Active Comparator): The arms of the study are just the order of the interventions are performed
  1. º Dry suction technique
  2. º Slow pull technique
  3. º Wet suction technique
  Interventions: Diagnostic Test: Dry suction technique (A); Diagnostic Test: Slow-pull technique (B); Diagnostic Test: Wet suction technique (C)
- ACB (Active Comparator): The arms of the study are just the order of the interventions are performed
  1. º Dry suction technique
  2. º Wet suction technique
  3. º Slow pull technique
  Interventions: Diagnostic Test: Dry suction technique (A); Diagnostic Test: Slow-pull technique (B); Diagnostic Test: Wet suction technique (C)
- BAC (Active Comparator): The arms of the study are just the order of the interventions are performed 2º Slow pull technique
  1º Dry suction technique 3º Wet suction technique
  Interventions: Diagnostic Test: Dry suction technique (A); Diagnostic Test: Slow-pull technique (B); Diagnostic Test: Wet suction technique (C)
- BCA (Active Comparator): The arms of the study are just the order of the interventions are performed
  1. º Slow pull technique
  2. º Wet suction technique
  3. º Dry suction technique
  Interventions: Diagnostic Test: Dry suction technique (A); Diagnostic Test: Slow-pull technique (B); Diagnostic Test: Wet suction technique (C)
- CAB (Active Comparator): The arms of the study are just the order of the interventions are performed
  1. º Wet suction technique
  2. º Dry suction technique
  3. º Slow pull technique
  Interventions: Diagnostic Test: Dry suction technique (A); Diagnostic Test: Slow-pull technique (B); Diagnostic Test: Wet suction technique (C)
- CBA (Active Comparator): The arms of the study are just the order of the interventions are performed
  1. º Wet suction technique
  2. º Slow pull technique
  3. º Dry suction technique
  Interventions: Diagnostic Test: Dry suction technique (A); Diagnostic Test: Slow-pull technique (B); Diagnostic Test: Wet suction technique (C)

INTERVENTIONS:
Diagnostic Test: Dry suction technique (A) — Using a linear echoendoscope, such as Pentax or Olympus, after identifying the lesion and deciding where to perform the EUS-FNB, always checking that there are no vessels on the eco-Doppler that would prevent puncture, a 22G Cook "Echo-Tip Procore" histology needle will be used to perform the following techniques of the described arms.
  - Dry suction puncture: Once the lesion is located and punctured, the stylet will be completely removed, and a 10 mL syringe with a vacuum of 10 mL will be attached. In each pass, the needle will be advanced and retracted 20-30 times according to the standard technique. The suction will then be closed, and the needle will be removed. The "fanning" technique will be performed whenever possible.
Diagnostic Test: Slow-pull technique (B) — Using a linear echoendoscope, such as Pentax or Olympus, after identifying the lesion and deciding where to perform the EUS-FNB, always checking that there are no vessels on the eco-Doppler that would prevent puncture, a 22G Cook "Echo-Tip Procore" histology needle will be used to perform the following techniques of the described arms.
Diagnostic Test: Wet suction technique (C) — Using a linear echoendoscope, such as Pentax or Olympus, after identifying the lesion and deciding where to perform the EUS-FNB, always checking that there are no vessels on the eco-Doppler that would prevent puncture, a 22G Cook "Echo-Tip Procore" histology needle will be used to perform the following techniques of the described arms.
  - Wet suction technique: Prior to puncture, the stylet should be removed and the needle should be flushed with 1-2 ml of physiological saline and a 10 ml vacuum syringe with 3-5 ml of saline should be attached. In each pass, the needle should be moved forward and backward 20-30 times. Aspiration should be opened as the needle advances and closed as it is withdrawn. Afterwards, the aspiration should be closed and the needle should be removed. The "fanning" technique should be performed whenever possible.

SUMMARY:
Endoscopic ultrasound (EUS) is a widely recognized tool for over 30 years for diagnosing intra-abdominal lesions and gastrointestinal cancers, especially pancreatic neoplasia. In most hospitals, it is the preferred method for sampling using fine-needle aspiration (EUS-FNA) or histology needle aspiration biopsy (EUS-FNB) to obtain cytological and histological material for an anatomopathological diagnosis. It is also recognized by current oncology guidelines.

Numerous factors can affect the efficacy of this technique, such as the needle size, type (cytology or histology), number of passes made on the lesion, the presence or absence of a pathologist in the endoscopy room, the experience of the endoscopist, etc.

Currently, EUS-FNA or EUS-FNB are recommended interchangeably for diagnosis; however, it appears that histology needles (EUS-FNB) allow for greater diagnostic efficacy by obtaining a cellular block with fewer passes, which allows for more advanced anatomopathological analysis (such as immunohistochemistry or molecular analysis).

Regarding the technique for performing the puncture and acquiring the sample, current European guidelines recommend sampling using EUS-FNA or FNB by dry suction with a 10 mL syringe. However, other recognized techniques, such as using a stylet with the "slow-pull" technique (not positioning for or against) or liquid biopsy (which could obtain larger cellular blocks compared to dry puncture), are widely used and could obtain better samples, but there is no clear consensus currently.

Investigators' goal is to conduct a randomized clinical trial of three EUS-FNB techniques (dry puncture vs slow-pull vs wet puncture) used in daily clinical practice to evaluate which of the three techniques has greater efficacy in cytological and pathological diagnosis.

ELIGIBILITY:
Inclusion criteria

* Age ≥ 18 years
* Patients referred for EUS-FNB after imaging tests (CT, MRI, or abdominal ultrasound) of pancreatic, non-pancreatic intraabdominal, mediastinal, or pelvic lesions greater than 1 cm.
* Signed informed consent.

Exclusion criteria

* Coagulopathy (INR> 1.5) or thrombocytopenia (<50,000)
* Severe heart or respiratory failure that contraindicates sedation.
* Use of anticoagulants and antiplatelet agents that cannot be suspended.
* Use of a needle of a different gauge to 22G
* Refusal to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2025-05-22 (Estimated); Study Completion 2025-05-22 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Efficacy | 2 years
  Analyze the diagnostic efficacy of the three techniques used in obtaining echoendoscopic biopsies of solid lesions: Slow-pull vs EUS-FNB with standard dry aspiration vs EUS-FNB with wet aspiration.
  The diagnostic efficacy will be evaluated in terms of sensibility, specificity, positive predictive value and negative predictive value.
Quality of samples | 2 years
  Tissue integrity A: presence of tissue cylinder (intact piece of tissue measuring at least 550 microns in the microscope field of view).B: presence of tissue cylinder that does not meet criteria but allows for a diagnosis based on cellular morphology.C: No viable intact tissue exists.Cellularity A: Satisfactory, presence of > 4 clusters suitable for cytological interpretation with a minimum of 10 cells.B: Adequate, presence of 2-4 clusters suitable for cytological interpretation with a minimum of 10 cells.C: Inadequate, < 2 clusters suitable for cytological interpretation or non-representative sample or a cell count < 50 with clear nuclear structures.Blood presence A: Minimal contamination, erythrocytes in < 25% B: Moderate contamination, erythrocytes in 25-50% C: Significant contamination, erythrocytes in > 50%

SECONDARY OUTCOMES:
Rapid On Site Evaluation (ROSE) | 2 years
  Impact of the presence of ROSE on the different EUS-FNB techniques
Endoscopist's experience | 2 years
  Evaluate the influence of the endoscopist's experience on the results of the three techniques. The experience of the endoscopic investigator will be based on the number of procedures divided in: more than 500 EUS-FNB, between 500-250 EUS-FNB and less than 250 EUS-FNB

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Perez-Aguado, MD, Principal Investigator — CHUIMI
Locations (2):
- Spain (2):
  - Hospital Universitario Doctor Negrin de Gran Canaria, Las Palmas de Gran Canaria, Las Palmas
  - Complejo Hospitalario Universitario Materno Infantil, Las Palmas de Gran Canaria, Las Palmas

IPD SHARING:
Plan to Share IPD: No